CLINICAL TRIAL: NCT05980403
Title: Prediction of Lymph Node Status in Stage T1 Esophageal Squamous Cell Carcinoma（RENMIN-237）
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yongshun Chen (Other)
Responsible Party: Sponsor-Investigator, Yongshun Chen, Professor, Renmin Hospital of Wuhan University
Organization: Renmin Hospital of Wuhan University (Other)
Other Study IDs: WDRY2023-K115
Record Dates: First submitted 2023-07-21; First posted 2023-08-08 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-01

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: superficial esophageal squamous cell carcinoma; lymph node metastasis; prediction model; tumor- infiltrating immune cells
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — tumor tissue samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Lymph node metastasis negative: Superficial esophageal squamous cell carcinoma with negative lymph node metastasis
- Lymph node metastasis positive: Superficial esophageal squamous cell carcinoma with positive lymph node metastasis
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention
  Groups: Lymph node metastasis positive

SUMMARY:
Accurate assessment of lymph node status in superficial esophageal squamous cell carcinoma is of great significance for preventing undertreatment and overtreatment. However, the accuracy of the commonly used preoperative imaging methods for evaluating lymph node status is not high, and it is urgent to develop a prediction model that can predict the risk of individual lymph node metastasis to assist in clinical decision-making. In this context, investigators intend to retrospectively collect the clinical and pathological data of 300 patients with superficial esophageal squamous cell carcinoma, construct a lymph node metastasis risk prediction model. In addition, investigators are also preparing to prospectively collect tissue samples from 30 patients with superficial esophageal squamous cell carcinoma to further explore the mechanism of lymph node metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with esophageal cancer in Renmin Hospital of Wuhan University from 2013 to 2022.
2. Histopathological diagnosis was squamous cell carcinoma.
3. T1NxM0.
4. Received endoscopic resection or esophagectomy.

Exclusion Criteria:

1. Patients who received neoadjuvant therapy.
2. Positive surgical margin.
3. Prior malignancy requiring active treatment within the previous 3 years except for locally curable cancers that have been apparently cured.
4. Lack of complete histopathological information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with superficial esophageal squamous cell carcinoma who underwent endoscopic therapy or esophagectomy.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-12-18 (Estimated)

PRIMARY OUTCOMES:
Lymphatic metastases | Through study completion, an average of 2 year
  The primary end point was the presence of lymph node metastases in surgically resected specimens (≥ 15 resected lymph nodes), or the development of metastases during follow-up including local recurrence and distant metastasis (AJCC 8th). In cases of an endoscopic resection prior to surgical resection, the tumor was found in the endoscopic resection specimen and lymph node status in the surgical resection specimen. When no additional surgery was performed after endoscopic resection, the development of metastases during follow-up was used as a surrogate end point.

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin hosptial of Wuhan University, Wuhan, Hubei, China